CLINICAL TRIAL: NCT01821729
Title: Phase II Feasibility Study of FOLFIRINOX-Losartan Followed by Accelerated Short Course Radiation Therapy With Capecitabine for Locally Advanced Pancreatic Cancer
Brief Title: Proton w/FOLFIRINOX-Losartan for Pancreatic Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Theodore Sunki Hong, Principal Investigator, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13-051
Record Dates: First submitted 2013-03-27; First posted 2013-04-01 (Estimated); Results first posted 2019-09-17 (Actual); Last update posted 2020-09-25 (Actual); Status verified 2020-09

CONDITIONS: Pancreatic Cancer
Keywords: Locally Advanced
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — folfirinox; Fluorouracil; Leucovorin; Oxaliplatin; Losartan; Proton Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Experimental Arm (Experimental): FOLFIRINOX, Losartan, Proton Beam Radiation Therapy
  Interventions: Drug: FOLFIRINOX; Drug: Losartan; Radiation: Proton Beam Radiation

INTERVENTIONS:
Drug: FOLFIRINOX — Oxaliplatin via IV on Day 1 over 2 hours; Irinotecan via IV on Day 1 over 90 minutes, 5FU via IV on Day 1 over 2-4 minutes
  Other Names: 5-Fluorouracil; 5FU; Leucovorin; Oxaliplatin
Drug: Losartan — Taken orally every day during Phase I for all 8 cycles
Radiation: Proton Beam Radiation — 30-45 minutes per day, daily Monday-Friday

SUMMARY:
This is a Phase II clinical trial, which tests the safety and effectiveness of an investigational combination of drugs to learn whether the combination of drugs works in treating a specific cancer. "Investigational" means that the combination of drugs is being studied. It also means that the FDA has not yet approved it for your type of cancer. Proton beam radiation therapy is an FDA approved radiation delivery system.

Conventional radiation therapy uses photons to treat cancer before patients undergo surgery to remove the tumor. In this study we are using radiation with protons, which spares surrounding tissue and organs from radiation. Proton radiation delivers radiation to the area requiring radiation with no dose beyond the treatment area. This may reduce side effects that patients would normally experience with conventional radiation therapy.

Researchers in the laboratory have discovered pathways inside cancer cells which contribute to the growth and survival of tumors. The FOLFIRINOX chemotherapy regimen is a combination of the drugs 5-fluorouracil, leucovorin and oxaliplatin. These chemotherapy drugs, along with the chemotherapy drug capecitabine, work by blocking these pathways and thereby preventing tumor growth. Capecitabine is FDA approved to be used alone or with other drugs to treat other types of advanced cancer, but not pancreatic cancer. In past research studies, FOLFIRINOX followed by radiation therapy with capecitabine has been identified as the most effective and active chemotherapy for patients with cancer that is spreading, and this is why we are using it to treat your type of cancer.

Losartan is classified as an angiotensin-receptor blocker (ARB), and is FDA approved for use in people with high blood pressure. Recent studies in people with different types of cancer, including pancreatic cancer, have shown that combining chemotherapy drugs with an ARB can help reduce/stop tumor growth more effectively than chemotherapy alone. Losartan has been used in previous research studies, and information from those research studies suggests that this drug in combination with FOLFIRINOX and capecitabine may be better at treating your type of cancer.

In this research study, we seek to determine whether combining FOLFIRINOX with Losartan before proton radiation therapy will be more efficient at controlling the growth of or shrinking your tumor than just FOLFIRINOX alone.

DETAILED DESCRIPTION:
If you are willing to participate in this research study, you will be asked to undergo some screening tests and procedures to confirm that you are eligible. Many of these tests and procedures are likely to be part of regular cancer care and may be done even if it turns out that you do not take part in the research study. If you have had some of these tests or procedures recently, they may or may not have to be repeated. These tests and procedures will include a medical history, routine physical exam, performance status, assessment of your tumor, routine blood tests, a blood sample to check your kidney function and a serum or urine pregnancy test if applicable. If these tests show that you are eligible to participate in the research study, you will begin the study treatment. If you do not meet the eligibility criteria, you will not be able to participate in this research study.

There are two phases to this study. Phase I involves FOLFIRINOX and Losartan. The treatment plant will begin with 8 cycles of FOLFIRINOX. Each cycle is 14 days, or 2 weeks long. FOLFIRINOX is comprised of four drugs: Oxaliplatin, irinotecan, fluorouracil and leucovorin. On Day 1 of each 14 day cycle, you will receive oxaliplatin via IV infusion over a period of 2 hours. Irinotecan will be administered via IV infusion on Day 1 of each cycle over a period of 90 minutes.

You will receive fluorouracil (5FU) on Day 1 of each cycle via IV infusion over a period of 2-4 minutes. You will then be fitted with an ambulatory infusion pump that will be delivered continuously over 46-48 hours.

In addition to these infusions, FOLFIRINOX will always be administered along with a two hours IV infusion of leucovorin, a drug composed of reduced folic acid, which helps enhance the effects of chemotherapy. You will be give leucovorin through a vein in your arm for 2 hours a day on Day 1 of each cycle.

You will also receive an injection of Neulasta after each FOLFIRINOX treatment. Neulasta is used to reduce the chance of infection from chemotherapy by boosting your white blood cell count. It will be administered 24-48 hours after your FOLFIRINOX infusion (on Day 3 or 4).

You will take one dose of Losartan by mouth every day during Phase I for all 8 cycles of FOLFIRINOX. If the dose of Losartan given to you during the first week does not give you any serious side effects, your dose will be increased once for the remainder of Phase I. We have provided a drug diary for you with instructions on how to take this tablet and what to do incase of any missed or vomited doses. We will monitor your response to treatment with a chest/abdominal CT after four cycles of FOLFIRINOX therapy (8 weeks).

Phase II involves Restaging/Proton Beam Radiation Therapy and Capecitabine. At this time your study doctor will assess for any progress in your cancer after the FOLFIRINOX + Losartan treatment again via CT scan. If your cancer has progressed, you will be removed from the study and continue with standard of care treatment. If it has not progressed, you will continue to the proton radiation therapy and capecitabine phase of the study.

During this phase you will receive proton beam radiation therapy at the Francis H. Burr Proton Therapy center for 1 week, Monday through Friday. Each visit is expected to take 30-45 minutes.

During the week of proton radiation therapy and for the week after, you will take capecitabine by mouth on Monday through Friday, for a total of ten days. You will be given a drug diary with instructions on how to take capecitabine and what to do in case of a missed or vomited dose.

You will receive the following tests and procedures at various time points during both portions of the study. These tests and procedures will include: routine blood tests, blood sample to check kidney function, CA19-9 and CEA blood tests, Chest CT/Abdominal-Pelvic CT, assessment for side effects, vital signs, performance status, routine physical exam and blood pressure monitoring.

After the final dose of study drug you will come into the clinic for follow-up visits for some assessments every 3 months until your cancer progresses. You will undergo the following tests: routine physical exam, vital signs, performance status, routine blood tests, assessment for side effects. In addition you are required to have a chest and abdominal/pelvic CT every 6 months for the first two years, and yearly for years 3-5. We would like to keep track of your medical condition for the rest of your life. We would like to do this by calling you on the telephone once a year to see how you are doing. Keeping in touch with you and checking on your condition every year helps us look at the long term effects of the research study.

ELIGIBILITY:
Inclusion Criteria:

* Cytologic or histologic proof pancreatic ductal carcinoma
* Locally advanced, unresectable disease
* Life expectancy of at least 3 months

Exclusion Criteria:

* Evidence of metastatic disease
* Pregnant or breastfeeding
* Serious concomitant systemic disorders incompatible with the study
* Already treated on ACE or ARB therapy for hypertension or renal protection at the time of enrollment
* Baseline hypotension
* Prior chemotherapy, radiation therapy, or biologic therapy for treatment of pancreatic tumor
* Treatment for other invasive carcinomas within the last 5 years who are greater than 5% risk of recurrence at the time of eligibility screening (carcinoma in-situ and basal cell carcinoma/squamous cell carcinoma of the skin are allowed)
* Other serious uncontrolled medical conditions
* Lack of physical integrity of the upper gastrointestinal tract or malabsorption syndrome
* Known, existing coagulopathy
* Prior systemic fluoropyrimidine therapy
* Participation in any investigational drug study within 4 weeks preceding the start of study treatment
* History of uncontrolled seizures, central nervous system disorders or psychiatric disability judged by the investigator to be clinically significant, precluding informed consent or interfering with compliance or oral drug intake
* Major surgery, excluding laparoscopy, within 4 weeks of the start of study treatment
* Taking cimetidine
* Receiving other study agents
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to 5-fluorouracil, irinotecan, oxaliplatin or losartan

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2013-07; Primary Completion 2018-07 (Actual); Study Completion 2021-09 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Theodore Hong, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Wang H, Yuan S, Wang H. Current Status of Research on Losartan in Tumour Therapy. J Cell Mol Med. 2026 Jan;30(1):e70985. doi: 10.1111/jcmm.70985. PMID 41486497
- [Derived] Murphy JE, Wo JY, Ryan DP, Clark JW, Jiang W, Yeap BY, Drapek LC, Ly L, Baglini CV, Blaszkowsky LS, Ferrone CR, Parikh AR, Weekes CD, Nipp RD, Kwak EL, Allen JN, Corcoran RB, Ting DT, Faris JE, Zhu AX, Goyal L, Berger DL, Qadan M, Lillemoe KD, Talele N, Jain RK, DeLaney TF, Duda DG, Boucher Y, Fernandez-Del Castillo C, Hong TS. Total Neoadjuvant Therapy With FOLFIRINOX in Combination With Losartan Followed by Chemoradiotherapy for Locally Advanced Pancreatic Cancer: A Phase 2 Clinical Trial. JAMA Oncol. 2019 Jul 1;5(7):1020-1027. doi: 10.1001/jamaoncol.2019.0892. PMID 31145418

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Experimental Arm
Started | 50
Received Chemoradiotherapy | 45
Underwent Attempted Surgery | 42
Completed | 49
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: Baseline characteristics are reported for all participants that started treatment. One participant withdrew consent prior to the start of study treatment.
Arm/Group | Experimental Arm
Number analyzed (Participants) | 49
Age, Continuous [Median (Full Range); unit: years] | 63 [42 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23
  Male | 26
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 49
ECOG PS [Count of Participants; unit: Participants] — Eastern Cooperative Oncology Group Performance Status: Lower scores indicate better functioning of daily activities of living. The score ranges from 0 to 5.
  Participants
    0 | 36
    1 | 13
CA19-9 level [Count of Participants; unit: Participants] — Carbohydrate antigen (CA) 19-9 is a type of antigen released by pancreatic cancer cells. Elevated CA 19-9 is associated with tumor growth.
  Participants
    <35 U/mL (Normal) | 9
    ≥ 35 U/mL (Elevated) | 40
CEA level [Count of Participants; unit: Participants] — Carcinoembryonic antigen is a bio-marker that is associated with some types of cancers. Elevated CEA levels can indicate the presence of a tumor. Population: CEA levels were not available for one participant
  Participants
    number analyzed (Participants) | 48
    <3.4 ng/mL (Normal) | 30
    ≥3.4 ng/mL (Elevated) | 18
Tumor site [Count of Participants; unit: Participants]
  Head | 31
  Body | 14
  Tail | 4
Tumor size [Median (Full Range); unit: mm] | 41 [18 to 68]
Vascular involvement [Count of Participants; unit: Participants] — Population: Two participants did not have vascular involvement
  Participants
    number analyzed (Participants) | 47
    Arterial alone | 15
    Venous alone | 11
    Arterial + venous | 21

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With R0 Resection
Description: The number of participants that received treatment with proton radiation along with FOLFIRINOX-Losartan and then subsequently underwent attempted surgery and achieved R0 resection. R0 resection means that no cancer cells were seen microscopically at the resection margin.
Time Frame: At the time of surgery (approximately 4 months after the start of treatment)
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental Arm
Number analyzed (Participants) | 49
Participants | 34

2. Secondary Outcome: Progression-Free Survival
Description: To determine the progression free survival of patients with locally advanced disease who receive FOLFIRINOX-Losartan and proton beam radiation therapy. Disease progression was assessed using Response Evaluation Criteria in Solid Tumors (RECIST 1.1).
  Progressive disease (PD): At least a 20% increase in the sum of the longest diameter (LD) of target lesion, taking as reference the smal lest sum LD recorded since the treatment started or the appearance of one or more new lesions (new lesions must be > slice thickness).
Time Frame: From the start of treatment until death or progression, median duration of 17.5 months
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Experimental Arm
Number analyzed (Participants) | 49
Months | 17.5 [13.9 to 22.7]

3. Secondary Outcome: Overall Survival for FOLFIRINOX + Proton Beam Radiation
Description: To determine overall survival in patients treated with preoperative FOLFIRINOX and proton beam radiation therapy
Time Frame: 2 years
Reporting Status: Not Posted

4. Secondary Outcome: Overall Survival for FOLFIRINOX Without Proton Radiation
Description: To determine the overall survival of patients with locally advanced disease who receive FOLFIRINOX-Losartan without proton radiation (i.e. patients who demonstrate progression at restaging)
Time Frame: 2 years
Reporting Status: Not Posted

5. Secondary Outcome: Determine Toxicity FOLFIRINOX-Losartan
Description: To determine the toxicity of FOLFIRINOX-Losartan in patients with locally advanced pancreatic disease
Time Frame: 2 years
Reporting Status: Not Posted

6. Secondary Outcome: Determine Toxicity of FOLFIRINOX-Losartan and Proton Beam Radiation
Description: To determine the toxicity of FOLFIRINOX-Losartan and proton beam radiation in patients with locally advanced pancreatic cancer.
Time Frame: 2 years
Reporting Status: Not Posted

7. Secondary Outcome: Rate of Downstaging
Description: To determine the rate of downstaging to surgical resection of FOLFIRINOX-Losartan followed by proton radiation in patients with locally advanced pancreatic cancer
Time Frame: 2 years
Reporting Status: Not Posted

8. Secondary Outcome: Determine Correlation of Somatic Gene Mutations and Outcome
Description: To determine the correlation between a panel of somatic genetic mutations (SNaPSHOT) and outcome in locally advanced pancreatic cancer treated with FOLFIRINOX-Losartan +/- proton beam radiation/capecitabine
Time Frame: 2 years
Reporting Status: Not Posted

9. Secondary Outcome: Determine Correlation Between Circulating Biomarkers and Outcome
Description: To determine the correlation between circulating biomarkers of TGF-B1 downregulation, including circulating Collagen I levels, and outcome in locally advanced pancreatic cancer treated with FOLFIRINOX-Losartan +/- proton beam radiation/capecitabine.
Time Frame: 2 years
Reporting Status: Not Posted

10. Secondary Outcome: Describe Quality of Life, Symptom Burden and Mood
Description: Describe quality of life, symptom burden and mood in the study population
Time Frame: 2 years
Reporting Status: Not Posted

11. Secondary Outcome: To Measure Utilization of Health Services
Description: To measure utilization of health services (ER, hospital and ICU visits) in the study population
Time Frame: 2 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: From the start of treatment until 30 days after the end of treatment, up to approximately 2 years
Arm/Group | Experimental Arm
All-Cause Mortality (participants affected / at risk) | 0/49
Serious Adverse Events (participants affected / at risk) | 15/49
Other Adverse Events (participants affected / at risk) | 40/49
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental Arm (N=49)
Anemia (Blood and lymphatic system disorders) | 2 (4)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1)
Fatigue (General disorders) | 2 (2)
General disorders and administration site conditions - Other, specify (General disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 2 (2)
Colitis (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 5 (6)
Mucositis oral (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 3 (4)
Vomiting (Gastrointestinal disorders) | 2 (3)
Alanine aminotransferase increased (Investigations) | 2 (3)
Aspartate aminotransferase increased (Investigations) | 1 (2)
Neutrophil count decreased (Investigations) | 5 (7)
Platelet count decreased (Investigations) | 3 (3)
Weight loss (Investigations) | 1 (1)
White blood cell decreased (Investigations) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 2 (2)
Ataxia (Nervous system disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental Arm (N=49)
Anemia (Blood and lymphatic system disorders) | 5 (11)
Cardiac disorders - Other, specify (Cardiac disorders) | 6 (8)
Chills (General disorders) | 6 (7)
Edema limbs (General disorders) | 10 (13)
Fatigue (General disorders) | 40 (124)
Fever (General disorders) | 10 (13)
Localized edema (General disorders) | 6 (7)
Malaise (General disorders) | 3 (3)
Non-cardiac chest pain (General disorders) | 3 (3)
Alopecia (Skin and subcutaneous tissue disorders) | 10 (14)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 3 (7)
Pruritus (Skin and subcutaneous tissue disorders) | 7 (11)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 13 (27)
Abdominal distension (Gastrointestinal disorders) | 9 (13)
Abdominal pain (Gastrointestinal disorders) | 37 (105)
Bloating (Gastrointestinal disorders) | 13 (16)
Colitis (Gastrointestinal disorders) | 3 (3)
Constipation (Gastrointestinal disorders) | 32 (72)
Diarrhea (Gastrointestinal disorders) | 29 (101)
Dry mouth (Gastrointestinal disorders) | 5 (7)
Dyspepsia (Gastrointestinal disorders) | 9 (13)
Dysphagia (Gastrointestinal disorders) | 7 (9)
Flatulence (Gastrointestinal disorders) | 13 (20)
Gastritis (Gastrointestinal disorders) | 3 (3)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 3 (3)
Hemorrhoidal hemorrhage (Gastrointestinal disorders) | 3 (4)
Malabsorption (Gastrointestinal disorders) | 11 (11)
Mucositis oral (Gastrointestinal disorders) | 12 (15)
Nausea (Gastrointestinal disorders) | 33 (123)
Oral pain (Gastrointestinal disorders) | 4 (4)
Vomiting (Gastrointestinal disorders) | 22 (53)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 13 (23)
Allergic reaction (Immune system disorders) | 5 (10)
Upper respiratory infection (Infections and infestations) | 3 (4)
Urinary tract infection (Infections and infestations) | 4 (4)
Infections and infestations - Other, specify (Infections and infestations) | 4 (6)
Bruising (Injury, poisoning and procedural complications) | 3 (3)
Alanine aminotransferase increased (Investigations) | 10 (14)
Aspartate aminotransferase increased (Investigations) | 5 (6)
Blood bilirubin increased (Investigations) | 9 (14)
Neutrophil count decreased (Investigations) | 6 (7)
Platelet count decreased (Investigations) | 13 (16)
Weight loss (Investigations) | 33 (91)
Anorexia (Metabolism and nutrition disorders) | 36 (80)
Dehydration (Metabolism and nutrition disorders) | 22 (59)
Hypokalemia (Metabolism and nutrition disorders) | 11 (21)
Hyponatremia (Metabolism and nutrition disorders) | 4 (5)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (6)
Back pain (Musculoskeletal and connective tissue disorders) | 19 (33)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 6 (8)
Myalgia (Musculoskeletal and connective tissue disorders) | 5 (5)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 (8)
Musculoskeletal and connective tissue disorder - (Musculoskeletal and connective tissue disorders) | 9 (20)
Concentration impairment (Nervous system disorders) | 4 (4)
Dizziness (Nervous system disorders) | 22 (37)
Dysarthria (Nervous system disorders) | 3 (3)
Dysgeusia (Nervous system disorders) | 18 (24)
Paresthesia (Nervous system disorders) | 4 (5)
Peripheral sensory neuropathy (Nervous system disorders) | 35 (131)
Spasticity (Nervous system disorders) | 3 (3)
Tremor (Nervous system disorders) | 3 (3)
Nervous system disorders - Other, specify (Nervous system disorders) | 9 (14)
Anxiety (Psychiatric disorders) | 22 (31)
Depression (Psychiatric disorders) | 7 (8)
Insomnia (Psychiatric disorders) | 20 (36)
Cough (Respiratory, thoracic and mediastinal disorders) | 6 (7)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 12 (15)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 8 (11)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 7 (7)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 4 (6)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 6 (8)
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 12 (24)
Hematuria (Renal and urinary disorders) | 3 (3)
Urinary frequency (Renal and urinary disorders) | 6 (8)
Urine discoloration (Renal and urinary disorders) | 3 (3)
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 3 (3)
Hypertension (Vascular disorders) | 3 (3)
Hypotension (Vascular disorders) | 16 (28)
Thromboembolic event (Vascular disorders) | 5 (5)
Vascular disorders - Other, specify (Vascular disorders) | 6 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-08-07): https://cdn.clinicaltrials.gov/large-docs/29/NCT01821729/Prot_SAP_000.pdf